CLINICAL TRIAL: NCT06879782
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Study on the Efficacy and Safety of Lifitegrast Ophthalmic Solution for the Treatment of Dry Eye Disease.
Brief Title: Phase III Clinical Study of Lifitegrast Ophthalmic Solution for the Treatment of Dry Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lunan Better Pharmaceutical Co., LTD. (Industry)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-LTST-ED-Ⅲ
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease (DED)
Keywords: Lifitegrast，Dry eye disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifitegrast (Experimental): Administer one drop of the ophthalmic solution in each eye, twice daily (morning and evening, approximately 12 hours apart), for a duration of 12 weeks.
  Interventions: Drug: Drug placebo
- placebo (Placebo Comparator): Administer one drop of the ophthalmic solution in each eye, twice daily (morning and evening, approximately 12 hours apart), for a duration of 12 weeks.
  Interventions: Drug: Drug placebo

INTERVENTIONS:
Drug: Drug placebo — Instill one drop of the eye solution in each eye, twice a day (morning and evening, approximately 12 hours apart), for a treatment period of 12 weeks.
  Other Names: Lifitegrast; Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical trial designed to evaluate the efficacy and safety of Lifitegrast Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signing of the informed consent form, willingness to comply with the treatment regimen prescribed by the trial protocol, and willingness to attend follow-up visits on time.
2. Age ≥18 years, regardless of gender.
3. Best corrected visual acuity ≥4.3 in both eyes (OU) at the screening visit (V1 visit).
4. History of dry eye disease in both eyes prior to the screening visit (V1 visit) (with at least one subjective symptom such as eye dryness, foreign body sensation, burning sensation, fatigue, discomfort, eye redness, or fluctuating vision).
5. Use of artificial tears within 30 days prior to the screening visit (V1 visit) to alleviate dry eye disease (DED) symptoms, with discontinuation of artificial tears at least 72 hours prior to the screening period, and willingness to refrain from using artificial tears during the trial.
6. Total Ocular Surface Disease Index (OSDI) score ≥13 at the screening visit (V1 visit).
7. Corneal fluorescein staining score ≥2 in at least one region of at least one eye and the same eye at both the screening visit (V1 visit) and baseline visit (V2 visit).
8. Conjunctival hyperemia score ≥1 in at least one eye at both V1 and V2 visits.
9. Eye Dryness Score (EDS) ≥40 (VAS score, OU) at both V1 and V2 visits.
10. At least one eye and the same eye meeting the following criteria at both V1 and V2 visits:

Inferior Corneal Fluorescein Staining Score (ICSS) ≥0.5; Schirmer's test (without anesthesia) ≥1 mm and ≤10 mm.- If both eyes meet the above criteria, the eye with the higher Inferior Corneal Fluorescein Staining Score (ICSS) at the V2 visit will be selected as the study eye. If both eyes have the same ICSS at the V2 visit, the eye with the lower Schirmer's Tear Test (STT) value at the V2 visit will be designated as the study eye. If both eyes have the same ICSS and STT values at the V2 visit, the right eye will be selected as the study eye.

Exclusion Criteria:

1. Currently suffering from ocular herpes or any other ocular infection or inflammation, or having a history of ocular herpes or any other ocular infection within 30 days prior to screening.
2. Presence of eyelid margin structural abnormalities (ectropion, entropion, eyelid laxity, etc.), severe conjunctivochalasis, Salzmann's nodular corneal degeneration, conjunctival goblet cell damage (e.g., vitamin A deficiency), progressive pterygium, wet age-related macular degeneration (wAMD), glaucoma, diabetic retinopathy, retinal vein occlusion, or other ocular diseases that, in the investigator's opinion, may increase the subject's risk or affect the trial results.
3. Ocular secondary scarring (e.g., radiation scars, chemical burns, Stevens-Johnson syndrome, cicatricial pemphigoid, etc.) that, in the investigator's opinion, may affect subject compliance or outcome assessment.
4. Subjects with secondary Sjögren's syndrome or other autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.), unless the subject meets the following conditions: a. Not using corticosteroids, immunomodulatory, or immunosuppressive drugs for the condition; b. The investigator considers that the medical condition will not affect the trial results.
5. History of organ or bone marrow transplantation.
6. Wearing contact lenses within 30 days prior to screening.
7. Undergoing physical treatments for dry eye (including eyelid scrubs, meibomian gland massage, warm compresses, steam treatments, etc.) within 30 days prior to screening.
8. Use of aspirin or aspirin-containing medications, non-steroidal drugs (including ocular or systemic use), or medications that may cause dry eye (e.g., anticholinergic drugs, serotonin reuptake inhibitors, etc.) within 30 days prior to the baseline visit (V2 visit), unless the subject has been on a stable dose for at least 30 days prior to the baseline visit and no change in dosage is expected during the trial.
9. Use of the following medications within the specified timeframes prior to the baseline visit (V2 visit): a. Ocular or systemic antihistamines, any ocular medications: within 14 days prior to V2 visit; b. Ocular cyclosporine, tacrolimus: within 6 weeks prior to V2 visit; c. Ocular or systemic corticosteroids, mast cell stabilizers: within 14 days prior to V2 visit.
10. History of punctal plug insertion or punctal cauterization within 12 weeks prior to screening.
11. Use of anti-glaucoma medications within 3 months prior to screening, history of non-laser glaucoma surgery, or laser glaucoma surgery within 6 months prior to screening.
12. History of YAG laser posterior capsulotomy within 6 months prior to screening, or corneal refractive surgery (e.g., LASIK) within 12 months prior to screening.
13. Known allergy to fluorescein, multiple allergies, or severe allergic diseases.
14. Presence of other uncontrolled clinical conditions (e.g., severe chronic infections, severe cardiopulmonary diseases, uncontrolled hypertension [defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg despite antihypertensive treatment], uncontrolled diabetes, malignancies, etc.).
15. Positive pregnancy test or lactating subjects (females only), or subjects of childbearing potential or male subjects with partners of childbearing potential who are unwilling to use contraception during the study and for 1 month after the last dose of study medication.
16. Participation in any other clinical trial involving investigational drugs/devices within 30 days prior to screening.
17. Poor compliance during the placebo washout period (compliance <80% or >120%).
18. Other conditions deemed unsuitable for enrollment by the investigator (e.g., depression, ocular mite infection, etc.). -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Inferior Corneal Fluorescein Staining Score | After 84 days of treatment
  After 84 days of treatment, the mean change from baseline in the Inferior Corneal Fluorescein Staining Score (ICSS，0-4) in the treatment group was compared with that in the placebo group. A higher corneal fluorescein staining score indicates a worse condition
Eye Dryness Score | After 84 days of treatment
  After 84 days of treatment, the mean change from baseline in the Eye Dryness Score (EDS, 0-100 [VAS, Visual Analog Scale]) in the treatment group was compared with that in the placebo group.A higher Eye Dryness Score indicates a worse condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China